CLINICAL TRIAL: NCT05087368
Title: An Observer-blinded, Randomized, Controlled, Phase 2 Study to Evaluate the Immunogenicity and Safety of Heterologous and Homologous Boosting With ChAdOx1-S and CoronaVac COVID-19 Vaccines or One Formulation of Clover Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2019) Determined in a lead-in Formulation Finding in Healthy Adults.
Brief Title: Immunogenicity and Safety of Heterologous and Homologous Boosting With ChAdOx1-S and CoronaVac or a Formulation of SCB-2019 (COVID-19)
Acronym: TP-SCB-2019001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Instituto Fernandes Figueira (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TP-SCB-2019-001
Record Dates: First submitted 2021-08-11; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Covid19
Keywords: Covid19; Immunogenicity; Vaccines
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Controlled, observer-blinded, Phase 2 Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be observer-blind for Stage 1 and Stage 2. The participants will be blinded before receiving the study vaccination. An unblinded dosing team, not involved with study participant's evaluation, will prepare and administer the study vaccines.
  The investigational product syringe will be opacified. The administration of the study vaccine will also be performed behind a closed curtain. The investigative study center personnel, as well as the sponsor personnel involved in the monitoring or conduct of the study, will be blinded to the study vaccine code.
  The laboratories will also be blinded, so that associating the sample with an assigned treatment or study visit will not be possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Stage 1 - Formulation-finding for SCB-2019 - Group 1 (Experimental): In Stage 1, immunogenicity and safety of three SCB-2019 formulations will be assessed in comparison with the ChAdOx1-S vaccine, in individuals who received two doses of ChAdOx1-S, 6 months (± 4 weeks) prior to recruitment.
  Participants (N=120) will be assigned to five groups for Stage 1 and receive doses as follows:
  Group 1: (N=30) Day 1: SCB-2019 (9 μg) alum;
  Interventions: Biological: Adjuvanted Recombinant SARS-CoV-2 TrimericS-protein Subunit Vaccine (SCB-2019 - Clover)
- Stage 1 - Formulation-finding for SCB-2019 - Group 2 (Experimental): In Stage 1, immunogenicity and safety of three SCB-2019 formulations will be assessed in comparison with the ChAdOx1-S vaccine, in individuals who received two doses of ChAdOx1-S, 6 months (± 4 weeks) prior to recruitment.
  Participants (N=120) will be assigned to five groups for Stage 1 and receive doses as follows:
  Group 2: (N=30) Day 1: SCB-2019 (9 μg) CpG 1018/alum;
  Interventions: Biological: Adjuvanted Recombinant SARS-CoV-2 TrimericS-protein Subunit Vaccine (SCB-2019 - Clover)
- Stage 1 - Formulation-finding for SCB-2019 - Group 3 (Experimental): In Stage 1, immunogenicity and safety of three SCB-2019 formulations will be assessed in comparison with the ChAdOx1-S vaccine, in individuals who received two doses of ChAdOx1-S, 6 months (± 4 weeks) prior to recruitment.
  Participants (N=120) will be assigned to five groups for Stage 1 and receive doses as follows:
  Group 3: (N=30) Day 1: SCB-2019 (30 μg) CpG 1018/alum;
  Interventions: Biological: Adjuvanted Recombinant SARS-CoV-2 TrimericS-protein Subunit Vaccine (SCB-2019 - Clover)
- Stage 1 - Formulation-finding for SCB-2019 - Group 4 (Experimental): In Stage 1, immunogenicity and safety of three SCB-2019 formulations will be assessed in comparison with the ChAdOx1-S vaccine, in individuals who received two doses of ChAdOx1-S, 6 months (± 4 weeks) prior to recruitment.
  Participants (N=120) will be assigned to five groups for Stage 1 and receive doses as follows:
  Group 4: (N=30) Day 1: ChAdOx1-S;
  Interventions: Biological: ChAdOx1-S COVID-19 Vaccine(Fiocruz/Oxford-AstraZeneca)
- Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 5 (Experimental): For Stage 2, immunogenicity of heterologous booster vaccination schedule (ChAdOx1-S (Group 5-7) - selected formulation of SCB-2019 or CoronaVac and CoronaVac (Group 8-10) - selected formulation of SCB-2019 or ChAdOx1) vs. a 2-dose ChAdOx1-S or CoronaVac series will be assessed.
  Participants (N=400) will be randomly (2:1:1) distributed into 6 groups for Stage 2 and receive doses as follows:
  Group 5: (N=100) Day 1 (boost) -SCB-2019;
  Interventions: Biological: Adjuvanted Recombinant SARS-CoV-2 TrimericS-protein Subunit Vaccine (SCB-2019 - Clover)
- Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 6 (Experimental): For Stage 2, immunogenicity of heterologous booster vaccination schedule (ChAdOx1-S (Group 5-7) - selected formulation of SCB-2019 or CoronaVac and CoronaVac (Group 8-10) - selected formulation of SCB-2019 or ChAdOx1) vs. a 2-dose ChAdOx1-S or CoronaVac series will be assessed.
  Participants (N=400) will be randomly (2:1:1) distributed into 6 groups for Stage 2 and receive doses as follows:
  Group 6: (N=50) Day 1 (boost) -ChAdOx1-S;
  Interventions: Biological: ChAdOx1-S COVID-19 Vaccine(Fiocruz/Oxford-AstraZeneca)
- Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 7 (Experimental): For Stage 2, immunogenicity of heterologous booster vaccination schedule (ChAdOx1-S (Group 5-7) - selected formulation of SCB-2019 or CoronaVac and CoronaVac (Group 8-10) - selected formulation of SCB-2019 or ChAdOx1) vs. a 2-dose ChAdOx1-S or CoronaVac series will be assessed.
  Participants (N=400) will be randomly (2:1:1) distributed into 6 groups for Stage 2 and receive doses as follows:
  Group 7: (N=50) Day 1 (boost) -CoronaVac;
  Interventions: Biological: CoronaVac (Sinovac Biotech)
- Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 8 (Experimental): For Stage 2, immunogenicity of heterologous booster vaccination schedule (ChAdOx1-S (Group 5-7) - selected formulation of SCB-2019 or CoronaVac and CoronaVac (Group 8-10) - selected formulation of SCB-2019 or ChAdOx1) vs. a 2-dose ChAdOx1-S or CoronaVac series will be assessed.
  Participants (N=400) will be randomly (2:1:1) distributed into 6 groups for Stage 2 and receive doses as follows:
  Group 8: (N=100) Day 1 (boost) -SCB-2019;
  Interventions: Biological: Adjuvanted Recombinant SARS-CoV-2 TrimericS-protein Subunit Vaccine (SCB-2019 - Clover)
- Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 9 (Experimental): For Stage 2, immunogenicity of heterologous booster vaccination schedule (ChAdOx1-S (Group 5-7) - selected formulation of SCB-2019 or CoronaVac and CoronaVac (Group 8-10) - selected formulation of SCB-2019 or ChAdOx1) vs. a 2-dose ChAdOx1-S or CoronaVac series will be assessed.
  Participants (N=400) will be randomly (2:1:1) distributed into 6 groups for Stage 2 and receive doses as follows:
  Group 9: (N=50) Day 1 (boost) - ChAdOx1-S;
  Interventions: Biological: ChAdOx1-S COVID-19 Vaccine(Fiocruz/Oxford-AstraZeneca)
- Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 10 (Experimental): For Stage 2, immunogenicity of heterologous booster vaccination schedule (ChAdOx1-S (Group 5-7) - selected formulation of SCB-2019 or CoronaVac and CoronaVac (Group 8-10) - selected formulation of SCB-2019 or ChAdOx1) vs. a 2-dose ChAdOx1-S or CoronaVac series will be assessed.
  Participants (N=400) will be randomly (2:1:1) distributed into 6 groups for Stage 2 and receive doses as follows:
  Group 10: (N=50) Day 1 (boost) - CoronaVac.
  Interventions: Biological: CoronaVac (Sinovac Biotech)

INTERVENTIONS:
Biological: ChAdOx1-S COVID-19 Vaccine(Fiocruz/Oxford-AstraZeneca) — Heterologous and Homologous Vaccination Series with ChAdOx1-S or CoronaVac COVID-19 Vaccines and Various Formulations of Clover Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2019) in Adults
  Arms: Stage 1 - Formulation-finding for SCB-2019 - Group 4; Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 6; Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 9
Biological: CoronaVac (Sinovac Biotech) — Heterologous and Homologous Vaccination Series with ChAdOx1-S or CoronaVac COVID-19 Vaccines and Various Formulations of Clover Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2019) in Adults
  Arms: Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 10; Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 7
Biological: Adjuvanted Recombinant SARS-CoV-2 TrimericS-protein Subunit Vaccine (SCB-2019 - Clover) — Heterologous and Homologous Vaccination Series with ChAdOx1-S or CoronaVac COVID-19 Vaccines and Various Formulations of Clover Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2019) in Adults
  Arms: Stage 1 - Formulation-finding for SCB-2019 - Group 1; Stage 1 - Formulation-finding for SCB-2019 - Group 2; Stage 1 - Formulation-finding for SCB-2019 - Group 3; Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 5; Stage 2 - Homologous vs. Heterologous Booster Regimen - Group 8

SUMMARY:
SARS-CoV-2 is a highly transmissible and pathogenic coronavirus that emerged in late 2019 and has caused a pandemic of acute respiratory disease, collectively called coronavirus disease-19 (COVID-19). SARS-CoV-2 has a high transmission rate, and severe cases of COVID-19 require admission to hospital intensive care units with the need for mechanical ventilation and associated high mortality. Currently cases continue to rise in many countries as the 'second and third waves' of SARS-CoV-2 infection evolve.

The authorized vaccines and most vaccines in development are focused on the major antigenic target of the virus, the SARS-CoV-2 spike (S) protein. Authorization was granted in Brazil by ANVISA for the Fiocruz/Oxford-AstraZeneca ChAdOx1-S COVID-19 vaccine as a 2-dose homologous vaccination regimen, 28- to 84-days apart. Emergency Use Authorization (EUA) was also granted for Sinovac Biotech's CoronaVac vaccine as a 2-dose homologous vaccination regimen, 28 days apart. Further vaccines, using different platforms are approved or expected to be approved for use against SARS-CoV-2. Most of the vaccines are expected to be authorized as 2-dose, homologous vaccination series.

SCB-2019 is Clover's adjuvanted recombinant SARS-CoV-2 trimeric S-protein subunit vaccine. The SCB-2019 antigen includes SARS-CoV-2 S protein as a trimer fused to Trimer-Tag and is produced in Chinese hamster ovary cells (CHO). SCB-2019 preserves the native trimeric structure of S-protein in the prefusion form and induces neutralizing antibodies to SARS-CoV-2. Trimer-Tag is derived from the fully-human C-propeptide domain of pro-collagen and is capable of self-trimerization, thus fusing any biologically-active proteins in-frame with Trimer-Tag. The resulting fusion proteins expressed in mammalian cells are secreted as disulfide bond-linked homotrimers.

The immunogenicity and safety of different dose levels (3, 9, and 30 μg) SCB-2019 vaccine, administered as 2-dose regimen 21-days apart was assessed in a phase 1 clinical study. All dose levels were well-tolerated and induced neutralizing antibodies against S protein of the SARS-CoV-2 virus. Based on the results of that study, Clover selected 30 μg of SCB-2019 in combination with the CpG 1018/alum adjuvant system for further evaluation in the phase 2/3 clinical program as having the most favorable benefit/risk profile. The pivotal study (CLO-SCB-2019-003) included approximately 30,000 healthy participants and individuals with stable pre-existing chronic medical conditions, is being conducted in multiple countries, including in Brazil. The primary purpose of that study (CLO-SCB-2019-003) is to demonstrate the safety and efficacy of SCB-2019 in the prevention of COVID-19. The study showed efficacy.

Heterologous boost vaccinations using different platforms may elicit immune responses of greater magnitude and breadth than can be achieved by priming or boosting with the same vaccine (He et al, 2021, Spencer et al., 2021). Also, given the anticipated challenges of vaccinating large proportions of the population, especially with respect to supply, out-of-stock situations, and potential misadministration, it is important for policy makers to have data on flexible vaccination schedules, where the third dose might be different from the priming platform. Protein-based adjuvanted vaccines have the advantage of being from a known and licensed technology that can produce high quantities of vaccine. Protein-based adjuvanted vaccines have also been shown to be highly immunogenic, both in the context of COVID-19 (Keech 2020; Richmond 2021) and other licensed vaccines (Skwarczynski 2016).

The purpose of this study is to compare the immunogenicity and safety of heterologous and homologous booster schedules in individuals who received ChAdOx1-S or CoronaVac vaccination previously. The study will be performed in 2 stages - Stage 1 will serve to down-select one of the SCB-2019 formulations for boosting. Stage 2 will compare homologous and heterologous booster regimens in individuals who have received a 2-dose primary vaccination series of either ChadOx1-S or of CoronaVac.

DETAILED DESCRIPTION:
This is a phase 2, randomized, controlled, observer-blinded, multi-center study to evaluate the immunogenicity and safety of heterologous and homologous vaccination series with ChAdOx1-S or CoronaVac COVID-19 vaccines and various formulations of adjuvanted recombinant SARS-CoV-2 trimeric S-protein subunit vaccine (SCB-2019). The study will be conducted in two stages.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Individuals are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests, and other study procedures.
3. Individuals are willing and able to give an informed consent, prior to screening.
4. Individuals who:

   • Received two dose of ChAdOx1-S vaccine 6 months (± 4 weeks) (Groups 1-4 of Stage 1 and Groups 5-7 of Stage 2) or CoronaVac 6 months (± 4 weeks) (Groups 8-10 of Stage 2) prior to recruitment in this study
5. Healthy participants or participants with pre-existing medical conditions who are in a stable medical condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
6. Female participants are eligible to participate in the study if not pregnant, not breastfeeding, and at least 1 of the following criteria apply:

   * Women of non-childbearing potential;
   * Women of childbearing potential (WOCBP) must have a negative urine pregnancy test prior to study vaccination. A confirmatory serum pregnancy test may be conducted at the investigator's discretion. They must be using a highly effective licensed method of birth control for 30 days prior to the first vaccination and must agree to continue such precautions during the study until 90 days after the last study vaccination.
7. Male participants must agree to employ acceptable contraception from the day of first dose of the study vaccine/comparator until 6 months after the last dose of the study vaccine/comparator and also refrain from donating sperm during this period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity - Stage 1 | Day 1
  Immunogenicity is defined as the ability of cells/tissues to provoke an immune response and is generally considered to be an undesirable physiological response, as measured by ELISA (homologous strain) and virus neutralization assay (homologous and heterologous strains).
Immunogenicity - Stage 1 | Day 15
  Immunogenicity is defined as the ability of cells/tissues to provoke an immune response and is generally considered to be an undesirable physiological response, as measured by ELISA (homologous strain) and virus neutralization assay (homologous and heterologous strains).
Immunogenicity - Stage 1 | Day 29
  Immunogenicity is defined as the ability of cells/tissues to provoke an immune response and is generally considered to be an undesirable physiological response, as measured by ELISA (homologous strain) and virus neutralization assay (homologous and heterologous strains).
Immunogenicity - Stage 2 | Day 1
  Immunogenicity is defined as the ability of cells/tissues to provoke an immune response and is generally considered to be an undesirable physiological response, as measured by ELISA (homologous strain) and virus neutralization assay (homologous and heterologous strains).
Immunogenicity - Stage 2 | Day 15
  Immunogenicity is defined as the ability of cells/tissues to provoke an immune response and is generally considered to be an undesirable physiological response, as measured by ELISA (homologous strain) and virus neutralization assay (homologous and heterologous strains).
Immunogenicity - Stage 2 | Day 180
  Immunogenicity is defined as the ability of cells/tissues to provoke an immune response and is generally considered to be an undesirable physiological response, as measured by ELISA (homologous strain) and virus neutralization assay (homologous and heterologous strains).
Immunogenicity - Stage 2 | Day 360
  Immunogenicity is defined as the ability of cells/tissues to provoke an immune response and is generally considered to be an undesirable physiological response, as measured by ELISA (homologous strain) and virus neutralization assay (homologous and heterologous strains).

SECONDARY OUTCOMES:
Reactogenicity | During 7 days after study vaccination
  Frequencies and percentages of participants experiencing local reactions and systemic solicited AEs; unsolicited AEs; SAEs; MAAEs and AESIs, will be summarized by vaccine group along with 95% CIs CI by the Clopper-Pearson method.
Reactogenicity | After 28 days after study vaccination
  Frequencies and percentages of participants experiencing local reactions and systemic solicited AEs; unsolicited AEs; SAEs; MAAEs and AESIs, will be summarized by vaccine group along with 95% CIs CI by the Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Ann Clemens Costa Clemens, MD, PhD, Study Director — Global Health - Oxford University Siena University
Locations (3):
- Brazil (3):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio de Grande Do Sul
  - Hospital Gloria D'or, Rio de Janeiro, Rio de
  - Centro de Estudos e Pesquisa em Moléstias Infecciosas (CEPCLIN), Natal, Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa Clemens SA, Milan EP, Sprinz E, Neto JC, Pacciarini F, Li P, Chen HL, Smolenov I, Pollard A, Clemens R. Homologous and Heterologous Boosting of the Chadox1-S1-S COVID-19 Vaccine With the SCB-2019 Vaccine Candidate: A Randomized, Controlled, Phase 2 Study. Open Forum Infect Dis. 2022 Aug 16;9(8):ofac418. doi: 10.1093/ofid/ofac418. eCollection 2022 Aug. PMID 36043184